CLINICAL TRIAL: NCT02922842
Title: A Study of Transcutaneous Electrical Nerve Stimulation for Overactive Bladder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: underenrollment
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: RSRB00060370
Record Dates: First submitted 2016-05-25; First posted 2016-10-04 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Urge Incontinence; Overactive Bladder
Keywords: transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Tibial Nerve (Active Comparator): Transcutaneous electrical stimulation will be placed on the posterior tibial nerve.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- Parasacral (Active Comparator): Transcutaneous electrical stimulation will be placed on the lower back near the s3 foramina.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- Shoulder (Sham Comparator): Transcutaneous electrical stimulation will be placed on the shoulder.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation
  Other Names: TENS device

SUMMARY:
The purpose of the study is to compare patient centered- outcomes between Transcutaneous Electrical Nerve Stimulation (TENS) at three locations to treat urinary urge incontinence. One of these locations will be along the tibial nerve, which is traditionally accessed near the medial malleolus. The second site will be on the sacral nerve which is accessed over the sacrum. The third site will be a sham site on the shoulder. This study will evaluate the feasibility of transcutaneous electrical stimulation in the treatment of overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are clinically diagnosed with urge incontinence, defined as urinary leakage associated with a sudden, strong desire to pass urine that is difficult to defer.
* Patients with urge predominant mixed incontinence.
* Patients will need to have answered at "Yes" to "leakage related to feeling urgency" on the UDI 6 questionnaire.
* Female
* Over 18 years of age.
* English speaking who are able to give informed consent to participate in the study.
* Patients who have four urinary incontinence episodes.

Exclusion Criteria:

* Stress incontinence desiring surgical management.
* Previous treatment of refractory urge incontinence such as PTNS, SNS, or Intradetrusor onabotulinumtoxin A injections.
* Neurological conditions affecting continence such as multiple sclerosis, a history of spinal shock within the past year, or neurologic impairment requiring a wheelchair.
* Urethral diverticulum.
* Daily catheterization due to urinary retention.
* The use of anticholinergic medications for less than 6 weeks.
* Patients who have pacemakers in place.
* Patients with limited mobility requiring a wheelchair.
* Elevated PVR > 200 cc
* Untreated urinary tract infection, defined as symptoms and a urine culture with greater than 100,000 cfu/ ml within the last 1 month prior to treatment.
* Uncorrected Stage 3 prolapse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07; Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Number of incontinence episodes per day | 6 weeks
  Patients will self-report the number of incontinence episodes.

SECONDARY OUTCOMES:
Number of bladder voids per day | 6 weeks
  Patients will self-report the number of times they void their bladder.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States